CLINICAL TRIAL: NCT00015054
Title: MPD04961-Methylphendidate Treatment of Cocaine Dependent ADHD Patients
Brief Title: Methylphendidate Treatment of Cocaine Dependent Patients With Attention Deficit Hyperactivity Disorder - 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Cincinnati MDRU (Other)
Masking: None | Purpose: Treatment
Other Study IDs: NIDA-5-0012-3; Y01-5-0012-3
Record Dates: First submitted 2001-04-18; First posted 2001-04-18 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 1999-02

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate

SUMMARY:
The purpose of this study is to demonstrate the feasibility of methylphenidate (MPD) as effective and safe in the outpatient treatment of cocaine-dependent patients with a comorbid DSM-IV diagnosis of Attention Deficit Hyperactivity Disorder (ADHD), to demonstrate the ability of each site to participate in a subsequent anticipated controlled trial of MPD (recruitment and execution), and to gather preliminary data on the ability of sweat patches to detect episodes of cocaine use.

DETAILED DESCRIPTION:
Forty-one participants were enrolled into this multi-site, outpatient, open-label, ten-week trial. Participants were scheduled to attend three visits per week to allow safety and efficacy measures to be taken. In addition, participants were given two hours of individual substance abuse therapy during the first four weeks, and one hour per week during the last six weeks, of the trial. All participants were started on a total daily dose of 20 mg MPD. The total daily dose was then increased to a maximum daily dose of 60 mg (20 mg TID) or to the maximum dose tolerated by the participant.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be between 21 and 50 years of age, male or female, of any race.
2. If female, subject cannot be pregnant or lactating.
3. Subject must be cocaine-dependent (as determined by the SCID and a clinical interview by a psychiatrist).
4. Subject must meet DSM-IV diagnostic criteria for ADHD:
5. Subject must have been actively using cocaine, (BE>300 ng/ml) within 30 days of the screening examination.
6. Subject must be negative for cocaine metabolites immediately prior to receiving a study treatment number and initial dose of MPD, as determined first by urine testing kit with result later confirmed by laboratory urine toxicology (BE < 300 ng/ml).
7. Subject must be willing and able to give informed consent.

Exclusion Criteria:

1. Subject has symptoms of AIDS.
2. Subject has a chronic medical disorder requiring medication.
3. Subject has a SCID Axis-I psychiatric diagnosis requiring medication.
4. Subject meets DSM-IV criteria for dependence for any substance except cocaine, alcohol, nicotine, marijuana, caffeine, and has been actively using during the past two weeks.
5. Subject is in need of detoxification from alcohol or benzodiazepines
6. Subject is taking psychotropic medication (except chloral hydrate for insomnia).
7. Subject is female of childbearing age who is at risk for becoming pregnant and is not using adequate contraceptive techniques as determined by the evaluating physician or Principal Investigator.
8. Subject has ALT or AST levels above three times laboratory normal
9. Subject has renal function tests (creatinine and BUN) or electrolyte levels (K, Na, Cl, HCO3) that are not within normal limits at baseline.
10. Subject has an EKG indicating clinically significant arrhythmias or abnormal conduction
11. Subject has organic brain syndrome (OBS) as evidenced in the psychiatric evaluation.
12. Subject has an acute or chronic medical or psychiatric condition which in the judgment of the evaluating physician would make study participation difficult or unsafe.
13. Subject has been enrolled in another research protocol within the past 45 days.
14. Subject has narrow angle glaucoma, by history
15. Subject has a diagnosis or family history of Tourettes syndrome
16. Subject has a history of seizures or seizure disorder
17. Subject has had an adverse reaction to methylphenidate
18. Subject has abnormal thyroid function (as determined by an abnormal T4 level that is clinically significant)
19. Subject has been treated for ADHD with psychomotor stimulants within the past month.
20. Subject plans to receive psychosocial treatment external to that designated in the protocol during study participation.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 1998-09; Primary Completion 1999-10 (Actual); Study Completion 1999-11 (Actual)

PRIMARY OUTCOMES:
Retention
Cocaine use
Global improvement

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Somoza, M.D., Ph.D., Principal Investigator — Cincinnati MDRU
Locations (1):
- Cincinnati MDRU, Cincinnati, Ohio, United States